CLINICAL TRIAL: NCT02110550
Title: Evaluation of IPS E.Max-CAD Endocrown in Molars Compared to the Conventional Design
Brief Title: Evaluation of a New Design of Crowns in the Posterior Teeth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UDDS-FixPro-01-2014
Record Dates: First submitted 2014-04-07; First posted 2014-04-10 (Estimated); Last update posted 2015-10-05 (Estimated); Status verified 2015-10

CONDITIONS: Broken Down Molars; IPS-emmax Crowns
Keywords: endocrown; marginal adaptation; anatomic form; retention loss; IPS.emmax crowns

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IPS.emmax crown (No Intervention)
- IPS.emmax endocrown (Experimental): Patients with excessively undermined and endodontically treated molars will receive the IPS.emmax endocrown as the restoration of choice.
  Interventions: Other: IPS.emmax endocrown

INTERVENTIONS:
Other: IPS.emmax endocrown
  Arms: IPS.emmax endocrown

SUMMARY:
Background: no randomized controlled trial has tried to compare treatment outcomes between the IPS.emmax endocrowns and the IPS.emmax conventional crowns .

Objective: to investigate the clinical performance of the IPS.emmax endocrowns and the IPS.emmax conventional crowns Design and setting: Parallel-groups randomized controlled trial on patients with one or more intensive damaged molars requiring crowning and being treated at the University of Damascus, Dental School in Damascus, Syria .All molars will be examined at the baseline assessment using a modified US Public Health Service (USPHS) criteria.

Participants: Incoming patients to the Fixed Prosthetic and Endodontic Departments will be examined to find any excessively damaged molars requiring crowning. Forty patients will be recruited according to specific inclusion criteria. Randomization will be performed using computer-generated tables; allocation will be concealed using sequentially numbered opaque and sealed envelopes.The included 40 patients will be analyzed (age range between 20-60 years). They will be randomly distributed into two groups with 20 patients in each group (1:1 allocation ratio).

Intervention: Excessively damaged and endodontically treated molars will be restored with IPS.emmax endocrowns or IPS.emmax crowns supported with composite core.

Main outcome measure: marginal adaptation and anatomic form will be investigated clinically and by apical radiographs at the baseline assessment using the modified (USPHS) at six assessment times during an 18-month observation period.

Assessor blinding will be employed.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 20 to 60 years old
* Good oral hygiene
* Gingival index (GI) equal 0
* Plaque index (PI) equal 0 or 1
* Primary acceptation and commitment to the trail

Inclusion criteria of molars:

* Two remaining axial walls at least.
* 0.5 mm above the gingival line at least for damaged axial walls.
* Good endodontic treatment and apical seal
* First and second upper and lower molars only.
* Against teeth could be natural or crowned.

Exclusion Criteria:

* Patients with an open bite or cross bite.
* Bruxism
* Periodontitis
* Gingival hyperplasia

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2014-05; Primary Completion 2015-09 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Change in Marginal Adaptation | at 3 months (T1), 6 months (T2), 9 months (T3), 12 months (T4), 15 months (T5), and 18 months (T6) following application
  The presence of marginal adaptation means that the restoration margins cannot be distinguished, the probe cannot find a step between the margins and the surrounding tissue, and no discoloration visible.
Change in the Anatomic Form | at 3 months (T1), 6 months (T2), 9 months (T3), 12 months (T4), 15 months (T5), and 18 months (T6) following application
  The anatomic form is considered satisfactory when the crown has a correct contour with tight proximal contact, no worn facets on restorations and no worn facets on opposing teeth.

SECONDARY OUTCOMES:
Change in the Retention Status | at 3 months (T1), 6 months (T2), 9 months (T3), 12 months (T4), 15 months (T5), and 18 months (T6) following application
  Retention loss is considered when the crown becomes loose or mobile.

CONTACTS AND LOCATIONS:
Overall Officials: Rana Dallool, DDS, Principal Investigator — University of Damascus Dental School
Locations (2):
- Syria (2):
  - Department of Fixed Prosthodontics, University of Damsacus, Damascus, Rif-dimashq Governorate
  - University of Damascus Dental School, Damascus, Rif-dimashq Governorate

REFERENCES:
- [Background] Bernhart J, Brauning A, Altenburger MJ, Wrbas KT. Cerec3D endocrowns--two-year clinical examination of CAD/CAM crowns for restoring endodontically treated molars. Int J Comput Dent. 2010;13(2):141-54. English, German. PMID 20648740
- [Background] Biacchi GR, Basting RT. Comparison of fracture strength of endocrowns and glass fiber post-retained conventional crowns. Oper Dent. 2012 Mar-Apr;37(2):130-6. doi: 10.2341/11-105-L. Epub 2011 Sep 26. PMID 21942234
- [Background] Bindl A, Mormann WH. Clinical evaluation of adhesively placed Cerec endo-crowns after 2 years--preliminary results. J Adhes Dent. 1999 Autumn;1(3):255-65. PMID 11725673
- [Background] Fischer H, Marx R. Fracture toughness of dental ceramics: comparison of bending and indentation method. Dent Mater. 2002 Jan;18(1):12-9. doi: 10.1016/s0109-5641(01)00005-7. PMID 11740960